CLINICAL TRIAL: NCT04250012
Title: Effectiveness of a Web-based Acceptance and Commitment Therapy for Wellbeing of Parents With Children With Chronic and Developmental Conditions: A Randomized Controlled Trial
Brief Title: Web-based ACT to Support Parents With Children With Chronic and Developmental Conditions
Acronym: Uupu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: The Gerocenter Foundation for Research and Development (Other); Social Insurance Institution, Finland (Other)
Responsible Party: Principal Investigator, Päivi Lappalainen, Principal Investigator, University of Jyvaskyla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/26/2018
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Burnout Syndrome; Psychological Distress; Depressive Symptoms; Quality of Life
Keywords: Parents, burnout, parental distress, Internet-based, ACT
MeSH Terms: conditions — Burnout, Psychological; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based ACT intervention (Experimental): Group "Internet-based ACT intervention" will receive a 10-week internet-based acceptance and commitment therapy intervention with three remote meetings with a psychologist
  Interventions: Behavioral: Internet-based ACT intervention
- Psychoeducation (Active Comparator): Group "Psychoeducation" will receive a self-help booklet and a link to mobile wellness training program
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Internet-based ACT intervention — The Internet-based ACT intervention included a 10-week web-based program consisting of five modules with different themes that the participants were instructed to process during the course of two weeks. The program was based on the processes of ACT and included themes such as life values, mindfulness, defusion, self-as-context acceptance and self-compassion. The content of each module consisted of text, video, exercises with audio files, and homework assignments. In addition, the participants filled in a diary with exercises in paper format. The intervention included also three remote meetings (à 45 minutes) via a videoconferencing tool doxy.me conducted by a psychologist. The remote meetings took place at the beginning, after 4 weeks, and at the end of the intervention.
  Arms: Internet-based ACT intervention
Behavioral: Psychoeducation — The psychoeducation group received a self-help booklet and a link to a web-based wellness training program. The program included exercises with MP3 audio files. No personal support during the 10-week intervention was provided.
  Arms: Psychoeducation

SUMMARY:
Parents of children with a chronic disease or functional disabilities have an increased risk of stress-related distress and reduced quality of life. Internet-delivered interventions are one way to reach out to exhausted parents who may often have challenges in finding time to access face-to-face services. We developed a guided web-based Acceptance and Commitment Therapy intervention for Finnish parents of children with chronic conditions or functional disabilities. Participants (N=100) will be recruited on parent associations' Facebook groups and randomly assigned to guided web-based ACT condition and a control condition receiving psychoeducation. The guided web-based ACT condition will receive a 10-week web intervention including three remote meetings with a psychologist through the telemedicine application Doxy.me. Symptoms of burnout (SMBQ), depression (PHQ), health-related quality of life (RAND-36), mindfulness (FFMQ), general measure of psychological flexibility (CompACT) as well as the wellbeing of their child (KINDL) will be measured before (pre) and after the intervention (post), at 7-month (follow-up 1) and 10-month (follow-up 2) after the pre-measurement. In this randomized controlled trial we will investigate the outcomes and the mechanisms of change of the web-based ACTintervention. In addition, we will examine the acceptability of the web-based intervention.

DETAILED DESCRIPTION:
Numerous studies have shown that parents of children with long-term and intellectual disabilities suffer more often from symptoms such as stress, anxiety and depression symptoms, feelings of uncertainty and fear, and loss of quality of life. In Finland, there are approximately 17.000 families where the illness or disability of a child under the age of 16 causes an extra daily burden for parents. Especially mothers of long-term or disabled children are vulnerable and have an increased risk of psychological symptoms. Parents of children with a chronic disease or functional disability also have an increased risk of stress-related distress and reduced quality of life. Prolonged psychological symptoms associated with caring for a child with a long-term illness can expose to chronic exhaustion and burnout, which can have serious health effects. The birth of a disabled child and the illness of a child with long-term illness also increases the risk of divorce in the family. Considering the hardship and challenges of this population group, special attention should be paid to their rehabilitation and access to services.

In Finland, for example, the Finnish Social Insurance Institution offers adaptation training and family-oriented rehabilitation courses for family caregivers. However, this form of support has limited availability and, on the other hand, is of relatively short duration. Several studies indicate, however, that the parents' mental health also affects the health and development of the child, and especially the long-term stress experienced by the parent can be harmful to children. The challenge is to motivate parents to take care of themselves and thus to have a better capacity to care for their children in need of special support. The majority of parents have a full-time employment, which also poses challenges for the forms of support. Therefore, the support of this parent group should focus on treatments that are easily available for them.

Web-based treatments offer one solution for delivering evidence-based psychological treatments for this distressed parents, who may often have challenges in finding time to access face-to-face services. Web-based interventions have been developed and tested for a wide range of health problems, including parental wellbeing. Advantages of web-based interventions are that they are not bound to time and place. They are available when most needed and enable integration of the intervention in everyday life.

Acceptance and commitment therapy (ACT) represents the third-wave of Cognitive Behavioral Therapies and incorporates mindfulness, experiential acceptance, and valued action (e.g., engagement in meaningful, values-driven activities) to promote psychological flexibility. Several studies and meta-analyses have shown that acceptance and commitment therapy has a positive effect on a variety of psychological symptoms. Promising results from web-based ACT interventions have been obtained for example for the treatment of stress, anxiety, and depression. ACT and other mindfulness-based treatments have been shown to improve psychological adjustment and to decrease stress in parents of children with developmental disabilities including autism and acquired brain injury.

The aim of the current study is to investigate the effectiveness of a web-based ACT intervention on wellbeing of parents with exhaustion and burnout symptoms, and whose children have chronic conditions and/or developmental disabilities. Effects will be investigated at before (pre) and after the intervention (post), at 7-month (follow-up 1) and 10-month (follow-up 2) after the pre-measurement. The research questions are the following:

1. Does the guided acceptance and commitment-based online intervention decrease the burnout and depression symptoms of parents of children with long-term illnesses and improve their quality of life, psychological flexibility, mindfulness skills, and cognitive strategies?
2. Which psychological processes (i.e., psychological flexibility, mindfulness skills, cognitive strategies) act as mediators of change?
3. Do the changes in the well-being of the parents improve the quality of life of the child?
4. How do parents experience online intervention and what kind of parent group especially will benefit from online support?

ELIGIBILITY:
Inclusion Criteria:

The parent:

* has a child (aged 0-18 years) with a long-term illness or developmental disorder or disability,
* has symptoms of burnout based on the Shirom-Melamed Burnout questionnaire (SMBQ), i.e. at least 2.75 points.
* has access to computer and internet.

Exclusion Criteria:

The parent:

* has an inadequate knowledge of the Finnish language (unable to fill in questionnaires or follow the program);
* has parallel regular psychological treatment or therapy
* has a severe mental disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Burnout | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  Burnout symptoms were measured with the Shirom-Melamed Burnout Questionnaire (SMBQ, Lundgren-Nilsson, Jonsdottir, Pallant, & Ahlborg, 2012; Melamed et al., 1999; Shirom & Melamed, 2006). The SMBQ measures four elements of burnout; Emotional exhaustion and physical fatigue, Listlessness, Tension, and Cognitive weariness. The SMBQ consists of 22 items that are rated on a seven-point scale ranging from 1 'Never or almost never' to 7 'Always or almost always'. High scores correspond to more burnout symptoms. The cut-off scores for burnout on the SMBQ are 2.75 - 3.74 indicating low burnout, 3,75 - 4,46 indicating high burnout and ≥ 4.47 indicating pathological level of burnout. SMBQ's psychometric characteristics and factorial validity have been supported (Lundgren-Nilsson et al., 2012; Shirom & Melamed, 2006).

SECONDARY OUTCOMES:
Depression (PHQ-9) | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  The PHQ-9 is one module of the larger Patient Health Questionnaire (Spitzer, Williams, & Kroenke, 2001), a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 comprises nine items that evaluate the presence of the nine Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (APA, 2000a) criteria for major depressive disorder in the previous 2 weeks. Each item of the PHQ-9 is rated on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day), for a total score ranging from 0 to 27. A final item assesses the perception of social, functional, and occupational impairment caused by the symptoms examined by the PHQ-9. Higher scores indicate an increased severity of depression symptoms .
Health-related quality of life (RAND-36) Health-related quality of life (RAND-36) Health-related quality of life (RAND-36) | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  The health-related quality of life (HRQL) will be measured with the Short-form 36 (SF-36), which is a validated and widely used generic quality of life questionnaire with good reliability. It consists of 36 questions measuring eight dimensions of quality of life: physical functioning, role functioning, pain, general health, vitality, social functioning, role functioning and mental health. Physical and mental component summary scores will be calculated. All 36 questions are scored on a scale from 0 to 100. Each scale is directly transformed into a 0-100 scale, with 100 representing the highest level of functioning possible. Lower scores indicate a worse outcome, i.e. more disability.
Mindfulness (FFMQ) | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  Mindfulness was assessed by the Five Facet Mindfulness Questionnaire (FFMQ, Baer et al., 2006). It includes 39-items that are rated on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true), with higher scores indicating higher levels of mindfulness skills. It includes the following elements. (a) Observing (b) Describing (c) Acting with awareness means (d) Non-judgment of inner experiences toward inner experiences. (e) Non-reactivity to inner experiences. The structure, reliability and validity of FFMQ have been supported (Baer et al., 2008).Higher scores indicate a better outcome, i.e. better mindfulness skills.
  Mindfulness was assessed by the Five Facet Mindfulness Questionnaire (FFMQ, Baer et al., 2006). It includes 39-items
Psychological flexibility and ACT-related processes (CompACT) | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  The Comprehensive Assessments of Acceptance and Commitment Therapy processes (CompACT; Francis et al., 2016) is a self-report questionnaire, with 23-items on a 7-points likert scale (0 = Strongly disagree, 6 = Strongly agree). The three-factor structure of the CompACT is concordant with recent accounts of psychological flexibility in terms of three dyadic processes; defined as: (1) openness to experience (acceptance; defusion); (2) behavioral awareness (present moment awareness; self as context); and (3) valued action (values; committed action). Higher scores in the full-scale (max 138 points) and on the subscales (Openness to experience, max 60 points, behavioral awareness, max 30 points, and valued action, max 48 points) indicate greater psychological flexibility, ie. a better outcome. These factors have demonstrated strong internal consistency.
Health-related quality of life in children (KINDL) | Change from baseline at 3 months, 7 months and 10 months after the pre-measurement
  The KINDL questionnaire is a generic instrument for assessing Health-Related Quality of Life in children and adolescents aged 3-17. There are three different versions of the instrument suitable for different age groups and developmental stages. Each version of the questionnaire can be completed both by children and adolescents, and also by their parents. The KINDL-questionnaire comprises twenty-four items yielding six dimensions (physical health, general health, family functioning, self-esteem, social functioning and school functioning) and a total score. The total score is transformed to a scale of 0-100 such that higher score represents a better outcome, i.e. better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Lappalainen, PhD, Study Director — Department of Psychology, University of Jyväskylä
Locations (1):
- Department of Psychology, University of Jyväskylä, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No